CLINICAL TRIAL: NCT02721433
Title: A Pragmatic Randomised, Multicentre Trial Comparing 4-weekly Versus 12-weekly Administration of Bone-targeted Agents in Patients With Bone Metastases From Either Castration-resistant Prostate Cancer or Breast Cancer - The REaCT-BTA Study
Brief Title: 4-weekly Versus 12-weekly Administration of Bone-targeted Agents in Patients With Bone Metastases
Acronym: REaCT-BTA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-01
Record Dates: First submitted 2016-03-10; First posted 2016-03-29 (Estimated); Last update posted 2020-12-02 (Actual); Status verified 2020-12

CONDITIONS: Breast Cancer; Prostate Cancer; Metastasis
MeSH Terms: conditions — Breast Neoplasms; Prostatic Neoplasms; Neoplasm Metastasis | interventions — Pamidronate; Denosumab; Zoledronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 4 weekly bone-targeted agent x 1 year (Active Comparator): Bone targeting agents as standard of care
  Interventions: Drug: Pamidronate; Drug: Denosumab; Drug: Zoledronate
- 12 weekly bone-targeted agent x 1 year (Active Comparator): Bone targeting agents as standard of care
  Interventions: Drug: Pamidronate; Drug: Denosumab; Drug: Zoledronate

INTERVENTIONS:
Drug: Pamidronate — Bone-targeted agent as standard of care
  Other Names: Aredia
Drug: Denosumab — Bone-targeted agent as standard of care
  Other Names: Prolia
Drug: Zoledronate — Bone-targeted agent as standard of care
  Other Names: Zometa

SUMMARY:
The current Rethinking Clinical Trials (REaCT) trial will compare two schedules(12- vs. 4-weekly) of bone-targeting agents (BTAs) to evaluate quality of life, pain and skeletal events within the Canadian Health Care System. This study will use an "integrated consent model" that involves "oral consent" rather than a written informed consent writing process as the study is comparing standard schedules and not a new administration schedule.

DETAILED DESCRIPTION:
Bone metastases are common in patients with advanced breast and prostate cancers. Skeletal metastases can be associated with reduced Quality of Life (QoL), pain and skeletal-related events (SREs) (defined as pathological fractures, surgery/radiotherapy to bone, spinal cord compression and hypercalcaemia). Maintaining QoL while avoiding or delaying SREs are the main goals of therapy. Patients therefore receive bone-targeted agents (e.g. pamidronate, zoledronate and denosumab) which are typically given every 4 weeks. However, this 4 week dosing is based on convenience so the treatment could be given concurrently with chemotherapy. The half-life of these drugs in the bone is many months or even years. Hence studies have been performed evaluating 12-weekly therapy. These have confirmed similar palliative outcomes in the 4 vs 12-weekly groups for both breast and prostate cancer patients. However, there remains clinical equipoise about which dosing interval physicians prescribe. The current trial will compare these two schedules of bone-targeting agents (12- vs. 4-weekly) to evaluate quality of life, pain and skeletal events within the Canadian Health Care System. This study will use an "integrated consent model" that involves "oral consent" rather than a written informed consent writing process as the study is comparing standard schedules and not a new administration schedule.

ELIGIBILITY:
Inclusion Criteria:

* Patients with either radiologically and/or histologically confirmed bone metastases from castrate resistant prostate cancer (36) or breast cancer.
* About to start or currently receiving BTA therapy.
* Serum creatinine >30 ml/min and corrected serum calcium ≥ 2 mmol/l
* Age ≥ 18 years.
* Able to provide verbal consent

Exclusion Criteria:

* For CRPC patients - Definite contraindication for denosumab at baseline (e.g. hypocalcaemia [Albumin-corrected serum calcium < 2.0 mmol/l]).
* History of or current evidence of osteonecrosis of the jaw.
* Radiotherapy or surgery to the bone planned within 4 weeks after randomization.
* Known hypersensitivity to trial drug or hypersensitivity to any other component of the trial drug (e.g. fructose).
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the trial protocol.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 263 (Actual)
Dates: Start 2016-08; Primary Completion 2019-09 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
Health related quality of life scores measured with European Organization for Research and Treatment of Cancer (EORTC) QLQ-C30 Functional Domain (Physical Subdomain) | 1 year
  Units on a scale

SECONDARY OUTCOMES:
Pain will be measured through the EORTC-Quality of Life Questionnaire (QLQ)-BM22 (pain domain) | 1 year
  Units on a scale
Health related quality of life scores | 1 year
  Units on a scale
Time to development of symptomatic skeletal events (SSEs) | 2 year
  SSEs defined from the date of randomization until the first date a patient experiences an SSE (an on-study SSE is defined as: use of radiotherapy to relieve skeletal symptoms, new symptomatic pathological bone fractures (vertebral or non-vertebral), spinal cord compression, tumour related orthopedic surgical intervention, hypercalcaemia). Any patient who does not experience a SSE will be censored on the last date the patient can be confirmed as SSE-free. Multiple measurements will be aggregated to arrive at one reported value.
Total number of and time to subsequent on study SSE - to calculate Skeletal Morbidity Rates | 2 year
  Multiple measurements will be aggregated to arrive at one reported value.
For sites where Edmonton Symptom Assessment Scores (ESAS) are performed as standard of care, the ESAS scores will also be collected. | 2 year
  Units on a scale
Adverse events/ toxicity profiles will be compared between the two different approaches. | 2 year
An economic analysis on Health Services Issues | 1 year
  We will perform a cost utility analysis alongside this pragmatic randomized controlled trial. The cost effectiveness of 4-week compared to 12-week BTA will be assessed in terms of the incremental cost per quality adjusted life year (QALY) gained from the perspective of health care system. Resource use and health utility will be measured from the trial at the follow up interviews. Health utility values would be estimated from the study questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Clemons, MD, Principal Investigator — The Ottawa Hospital
Locations (1):
- The Ottawa Hospital Research Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available.

REFERENCES:
- [Derived] Tu MM, Clemons M, Stober C, Jeong A, Vandermeer L, Mates M, Blanchette P, Joy AA, Aseyev O, Pond G, Fergusson D, Ng TL, Thavorn K. Cost-Effectiveness Analysis of 12-Versus 4-Weekly Administration of Bone-Targeted Agents in Patients with Bone Metastases from Breast and Castration-Resistant Prostate Cancer. Curr Oncol. 2021 May 13;28(3):1847-1856. doi: 10.3390/curroncol28030171. PMID 34068083